CLINICAL TRIAL: NCT05914532
Title: In Patients With Axial Spondyloarthropathy; Evaluation of the Relationship Between the Systemic Immune Inflammation Index and the Systemic Inflammatory Response Index With Disease Activity and Function
Brief Title: New Biomarkers in Axial Sypondyloarthropathy; SII and SIRI
Status: Completed | Type: Observational
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Burak Tayyip Dede, Physical Medicine and Rehabilitation, Istanbul Training and Research Hospital
Other Study IDs: 19/08/2022, 2011-KAEK-50: 262
Record Dates: First submitted 2023-06-10; First posted 2023-06-22 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Axial Spondyloarthritis
Keywords: Axial Spondyloarthritis; Systemic Immune Inflammation Index; Systemic Inflammation Response Index
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: healthy controls
  Interventions: Other: lab testing
- group 2: axial spondyloarthropathy
  Interventions: Other: lab testing

INTERVENTIONS:
Other: lab testing — Complete blood count and erythrocyte sedimentation rate and C-reactive protein values of the participants were analyzed by laboratory test.

SUMMARY:
investigators aimed to evaluate the relationship between Systemic Immune Inflammation Index (SII) and Systemic Inflammation Response Index (SIRI) and disease activity in patients with axial spondyloarthropathy (SpA).

DETAILED DESCRIPTION:
The clinical characteristics and laboratory data of the patients and healthy controls participating in our study were obtained through the hospital system. Then, the new biomarkers SIRI and SII values were calculated. SIRI= neutrophil count*monocyte count/lymphocyte count and SII= neutrophil count*platelet count/lymphocyte count. Then, SIRI and SII values were compared between groups. The relationship between disease activity and SIRI and SII values in the patient group was examined.

ELIGIBILITY:
Inclusion Criteria:

* SpA patients diagnosed according to the 2009 Assessment of Spondyloarthritis International Society classification criteria
* 51 healthy controls working in our hospital,

Exclusion Criteria:

infections, coronary artery disease, kidney and liver dysfunction, cancer diagnosis, surgery in the last three months, diabetes mellitus diagnosis, hypertension and pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1:healthy controls working in our hospital,
  Group 2: SpA patients diagnosed according to the 2009 Assessment of Spondyloarthritis International Society classification criteria
Sampling Method: Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Comparison of SIRI and SII between Patient and Healthy Control | Baseline
  SIRI= neutrophil count*monocyte count/lymphocyte count and SII= neutrophil count*platelet count/lymphocyte count.

SECONDARY OUTCOMES:
Correlation analysis of SIRI and SII with scales and laboratory findings | Baseline
  SIRI= neutrophil count*monocyte count/lymphocyte count and SII= neutrophil count*platelet count/lymphocyte count.

CONTACTS AND LOCATIONS:
Overall Officials: Burak Tayyip DEDE, MD, Principal Investigator — İstanbul Training and Research Hospital
Locations (1):
- Istanbul Training and Resarch Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu J, Yan L, Chai K. Systemic immune-inflammation index is associated with disease activity in patients with ankylosing spondylitis. J Clin Lab Anal. 2021 Sep;35(9):e23964. doi: 10.1002/jcla.23964. Epub 2021 Aug 21. PMID 34418163